CLINICAL TRIAL: NCT02864719
Title: An Intervention for Cardiac Arrest Survivors With Chronic Fatigue: A Feasibility Study
Brief Title: An Intervention for Cardiac Arrest Survivors With Chronic Fatigue
Acronym: CAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Young J Kim, Research associate, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO09110375
Record Dates: First submitted 2016-05-06; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Heart Arrest; Cardiac Arrest; Fatigue
Keywords: Heart arrest; Cardiac arrest; Fatigue
MeSH Terms: conditions — Heart Arrest; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Energy Conservation+Problem Solving Therapy (Experimental): The intervention was delivered by telephone. Each EC+PST intervention session was planned to last approximately 45 minutes and occur twice a week for up to 4 weeks. Sessions terminated when the participants identified and solved two fatigue-related problems of their choice or had participated in the intervention for eight sessions. A Participant Workbook was used throughout the intervention. During eight intervention sessions, participants identified two fatigue-related problems and solutions for them, implemented the solution plans, and reviewed the implementations.
  Interventions: Other: Energy Conservation+Problem Solving Therapy

INTERVENTIONS:
Other: Energy Conservation+Problem Solving Therapy — The intervention was delivered by telephone. Each EC+PST intervention session was planned to last approximately 45 minutes and occur twice a week for up to 4 weeks. Sessions terminated when the participants identified and solved two fatigue-related problems of their choice or had participated in the intervention for eight sessions. A Participant Workbook was used throughout the intervention. During eight intervention sessions, participants identified two fatigue-related problems and solutions for them, implemented the solution plans, and reviewed the implementations.

SUMMARY:
The primary aim was to examine the feasibility of an Energy Conservation + Problem Solving Therapy (EC+PST) intervention delivered over the telephone and to evaluate the preliminary intervention effect on fatigue impact in daily activities in post-cardiac arrest (CA) adults with chronic fatigue.

DETAILED DESCRIPTION:
The primary aim was to examine the feasibility of recruiting and retaining participants for an Energy Conservation + Problem Solving Therapy (EC+PST) intervention delivered over the telephone, to evaluate the acceptability of the intervention, and to assess the appropriateness of the outcome measures. The secondary aim was to evaluate the preliminary intervention effect on fatigue impact, activity performance, and participation in daily activities in post-cardiac arrest (CA) adults with chronic fatigue.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months post-cardiac arrest
* Presence of moderate-to-severe fatigue: ≥ 4 score on the Fatigue Severity Scale
* Availability of landline telephone or cell phone
* Living within 150 miles of the University of Pittsburgh, Oakland
* Functional English fluency and literacy
* Intact cognition
* Community living

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of people who completed their study participation | Week 5
  Assessing the feasibility of recruitment and retention
Number of participants who successfully identified and solved fatigue-related problems | Week 5
  Assessing the feasibility of telephone intervention delivery
Client Satisfaction Questionnaire - 8 | Week 5
  * Assessing the participants' satisfaction and the acceptability of the intervention
  * Four-point scale ranging from 1 to 4, and a total score ranging from 8 - 32 with higher scores indicating greater satisfaction
Understanding of Materials Scale | Week 5
  * Assessing the clarity of the Participant Workbook and the acceptability of the intervention
  * Five-point scale ranging from 1 (strongly disagree) to 5 (strongly agree), and a total score ranging from 0 to 50, with higher scores indicating greater understanding of the workbook

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale | Week 0 and Week 5
  * Assessing how fatigue has impacted performance in functional activities
  * 21 items in three subscales with scores ranging from 0 to 84: physical, cognitive, and psychosocial subscales. The higher the total scores, the greater the impact of fatigue
Fatigue Severity Scale | Week 0 and Week 5
  * Measuring the severity of fatigue by self-report
  * Total score is the mean of scores ranging from 1 to 7, and a higher score indicates having more severe fatigue.
Patient-Reported Outcomes Measurement Information System Fatigue Scale | Week 0 and Week 5
  * Measuring overall fatigue by self-report and computerized adaptive test
  * Total score ranging from 10 to 90 with the average score of the US general population is 50. The higher the total score, the worse the fatigue.
Performance Assessment of Self-Care Skills - Self-report (PASS-SR) | Week 0 and Week 5
  * Measuring perceived performance in activities of daily living by self-report
  * The total mean scores (habit and skill separately) ranging from 3 to 0, and the higher mean score indicates less difficulty in performing activities of daily living
Functional Activities Questionnaire | Week 0 and Week 5
  * Measuring perceived performance in higher level instrumental activities of daily living by self-report
  * A total score ranging from 0 to 30, and a higher total score indicates having more difficulty performing daily activities
Participation Objective, Participation Subjective (POPS) | Week 0 and Week 5
  * Measuring participation in activities of daily living by self-report
  * Participation Objective sub-scale score ranges from -3 (the least proportion, frequency, or hours) to +3 (the greatest proportion, frequency, or hours); Participation Subjective sub-scale score ranges from -4 (participating in the most important area, but wanting to engage either more or less) to +4 (participating in the most important area with satisfaction).